CLINICAL TRIAL: NCT01706406
Title: Group Psychoeducational Treatment for Women With Sexual Arousal Difficulties, Phase II
Acronym: Group PED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Lori Brotto, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C05-0400-II
Record Dates: First submitted 2010-10-29; First posted 2012-10-15 (Estimated); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Low Female Sexual Arousal; Low Female Sexual Desire
Keywords: female sexual arousal; female sexual desire; psychoeducational intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 treatment (Experimental): Women randomized into the "treatment" group will undergo pre-treatment testing (questionnaires and physiological assessment)within 14 days of beginning treatment
  Interventions: Behavioral: Brief psychoeducational intervention for female sexual arousal disorder
- 2 waitlist (Other): Women randomized to the "waitlist" group will undergo initial testing (questionnaires and physiological testing) and receive no treatment until the next scheduled group (4 months). They will undergo pretreatment testing and treatment on the same schedule as women in the "treatment" group.
  Interventions: Behavioral: Brief psychoeducational intervention for female sexual arousal disorder

INTERVENTIONS:
Behavioral: Brief psychoeducational intervention for female sexual arousal disorder — four 1.5 hour long group psychoeducational sessions, spaced 2 weeks apart for a total of 8 weeks.

SUMMARY:
The purpose of this study is to pilot test and determine the efficacy of a psychoeducational intervention (PED) we recently piloted in a group format for women with acquired sexual arousal disorder (FSAD).

HYPOTHESES:

1. - Compared to baseline measures, the PED will result in significant improvement in self-report measures of: (a) subjective sexual arousal; (b) perception of genital arousal/genital sensitivity; (c) orgasmic experience; (d) sexual desire; (e) sexual distress; (f) relationship satisfaction; (g) depressive symptoms; and (h) quality of life.
2. - It is unknown what effect the PED will have on actual physiological sexual arousal.
3. - The group format will be a feasible and cost-effective method of delivering empirically supported treatment to women with sexual arousal difficulties and will contribute towards meeting the needs for sexual health care for women on the clinic wait-list at the BC Centre for Sexual Medicine.

DETAILED DESCRIPTION:
Sexual arousal difficulties are common among women, affecting approximately 22% of women between the ages of 18 and 59 (Laumann, Paik & Rosen, 1999). Although there are evidence-based psychological treatments available for women with orgasmic and pain disorders, there are currently no empirically-supported treatments for women with acquired Sexual Arousal Disorder (FSAD). Moreover, there have been numerous attempts to find evidence for a pharmacological agent effective at treating women's sexual arousal complaints; however, to date these studies have been inconclusive. Given the significant role that sexual health plays in quality of life, the fact that effective psychological treatments for women's sexual dysfunction are not widely available, and the fact that wait-lists to see health care professionals with expertise in the area of sexual dysfunction are often unwieldy, there is a need to establish brief, evidence-based approaches to treat women's acquired FSAD. Psychological therapy in a group format is a standard practice at the BC Centre for Sexual Medicine. However, in this study we would like to collect information from participants that would help us in determining the specific efficacy of the PED as well as identifying demographic or participant variables that might predict a positive response to the PED. Because we are using this information to determine the treatment's efficacy and because we will use this information as the basis for a publication, we deem this to be a research trial in which ethics review is necessary.

OBJECTIVES: We have recently developed and tested a new psychoeducational treatment (PED) for the treatment of FSAD due to early-stage gynecologic cancer treatment, and for healthy women with FSAD. Our data show this PED to significantly improve self-reported sexual desire, arousal, mood, relationship distress, and quality of life. We are currently testing the efficacy of this PED in a larger sample of cancer survivors with FSAD. The goal for this study is to determine the efficacy of the group PED for currently seeking treatment at the BC Centre for Sexual Medicine for FSAD. By using a waitlist control group, we can determine if any improvement in sexual function is due to treatment or the passage of time.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 19 and 65
* currently seeking treatment at the BC Centre for Sexual Medicine
* meet clinical criteria for acquired Female Sexual Arousal Disorder (FSAD);
* be proficient in English and willing to take part in group sessions.

Exclusion Criteria:

* does not meet clinical criteria for acquired Female Sexual Arousal Disorder (FSAD)
* not currently Seeking seeking treatment at the BC Centre for Sexual Medicine

Ages: 19 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2007-11; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Change in physiological sexual arousal | Sexual arousal will be measured approximately one week pre-treatment and approxiately two weeks post-treatment
  Sexual arousal will be measured physiologically with a Vaginal Photoplethysmograph (VPP). The VPP measures vaginal pulse amplitude (VPA) which has been found to be a sensitive and specific measure of genital arousal (Laan & Everaerd, 1995).
Long-term change in physiological sexual arousal | Sexual arousal will be assessed approximately one-week pre-treatment and approximately 6 months post treatment
  Sexual arousal will be measured physiologically with a Vaginal Photoplethysmograph (VPP). The VPP measures vaginal pulse amplitude (VPA) which has been found to be a sensitive and specific measure of genital arousal (Laan & Everaerd, 1995).

SECONDARY OUTCOMES:
Subjective sexual arousal | Subjective sexual arousal will be assessed approximately one week pre-treatment, approximately two-weeks post-treatment and approximately 6-months post treatment
  The Female Sexual Function Inventory (FSFI; Rosen et al. 2000) questionnaire will be used to measure subjective sexual arousal. The FSFI a 19-item self-report questionnaire which assesses sexual function in women. It covers six sexual domains: lubrication, arousal, desire, pain, orgasm and satisfaction.

OTHER OUTCOMES:
Sexual Distress | Sexual distress will be assessed approximately one week pre-treatment, approximatley two weeks post-treatment and approximately 6-months post-treatment
  Sexual distress will be measured with the Female Sexual Distress Scale (FSDS, Derogatis et al. 2002). The FSDS is a 12-item self-report questionnaire assessing for sexuality related personal distress.
Mood | Mood will be assessed approximately one week pre-treatment, approximatley two weeks post-treatment and approximately 6-months post-treatment
  Mood will be measured with the Beck Depression Inventory (BDI; Beck & Beamesderfer, 1974), a widely-used self-report questionnaire designed to assess the severity of depressive symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Lori A Brotto, PhD, Principal Investigator — University of British Columbia
Locations (2):
- Canada (2):
  - BC Centre for Sexual Medicine, Vancouver, British Columbia
  - UBC Sexual Health Lab, Vancouver Hospital, Vancouver, British Columbia

REFERENCES:
- See also: UBC Sexual Health Lab website — http://www.obgyn.ubc.ca/SexualHealth